CLINICAL TRIAL: NCT03944291
Title: Unilateral vs. Bilateral Pudendal Nerve Block for Post-Episiotomy Pain Relief: A Randomized Clinical Trial
Brief Title: Pudendal Nerve Block for Post-Episiotomy Pain Relief
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AS1871
Record Dates: First submitted 2019-05-08; First posted 2019-05-09 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Intervention Model Description: Bupivacaine
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unilateral PNB (Active Comparator): Unilateral Pudendal Nerve Block
  Interventions: Procedure: Pudendal Nerve Block
- Bilateral PNB (Active Comparator): Bilateral Pudendal Nerve Block
  Interventions: Procedure: Pudendal Nerve Block

INTERVENTIONS:
Procedure: Pudendal Nerve Block — Pudendal Nerve Block
  Other Names: Bupivacaine

SUMMARY:
Unilateral vs. Bilateral Pudendal Nerve Block for Post-Episiotomy Pain Relief: A Randomized Clinical Trial

ELIGIBILITY:
Inclusion Criteria:

* Term (37 to 42 weeks gestation), primigravid women with singleton vertex fetus

Exclusion Criteria:

* Women with bleeding disorders, known hypersensitivity to local anesthetics, chronic use of pain medication, had previous vaginal surgery, extensive vulvovaginal infection, malposition or malpresentation were excluded from the study. Also, women who failed to deliver vaginally, had extensive perineal or cervicat tears, or had instrumental delivery were excluded from the final analysis of the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale for pain scoring | 48 hours
  visual analogue scale (VAS) from 0 to 100 with 0 corresponding to no pain at all and 100 as the worst pain the woman can describe

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt